CLINICAL TRIAL: NCT01968902
Title: A Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Incobotulinumtoxin Type A for the Functional Improvement of Lower Extremity Spasticity in Patients With Multiple Sclerosis
Brief Title: Safety of Xeomin for Lower Limb Spasticity in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Multiple Sclerosis Center of Northeastern New York (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPASTICITY-001
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Muscle Spasticity; Multiple Sclerosis
Keywords: spasticity; lower limb; multiple sclerosis; toxin
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- incabotulinumtoxinA (Active Comparator): intramuscular injection, 200 to 400 units, 1 injection visit only
  Interventions: Biological: incabotulinumtoxinA
- Placebo (Placebo Comparator): intramuscular injection, saline 200 - 400 units , 1 injection visit only
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: incabotulinumtoxinA — A dose of 200 units to 400 units of Xeomin will be injected by EMG-guided technique into the appropriate muscles in the effected leg at injection visit
  Other Names: Xeomin®
  Arms: incabotulinumtoxinA
Biological: Placebo — Saline injection on the day of injection visit
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Xeomin® will prove effective for significantly improving lower extremity spasticity and will be well tolerated by the majority of MS patients.

DETAILED DESCRIPTION:
Overall Design: Thirty patients with MS, male or female, ages 18-70, either relapsing or progressive types, are to be evaluated in a prospective treatment trial comparing gait before and after injections of Xeomin.

Patient Population: The patients included are to have functionally significant equinovarus spasticity in primarily one lower extremity; functionally significant spasticity is defined as spasticity impairing gait during observation of during a 25 foot walk, causing falls, or leading to secondary orthopedic complications such as genu recurvatum or pain in the low back or hip. The patients are to be ambulatory, with stable disease.

Dose Selection: A dose of 200 units to 400 units of Xeomin will be injected by EMG-guided technique into the appropriate muscles in the effected leg. These muscles may include gastrocnemius and soleus, tibialis posterior or other muscles as determined by the examiner. The dose administered will be determined by the blinded injector based on determination of muscle bulk and the degree of spasticity Blinding: Investigators will be blinded to medication used throughout study. Site will randomize subjects in a 1:1 fashion by using an unblinded site delegate.

Compliance with Laws and Regulations: This study will be conducted in accordance with the U.S. Food and Drug Administration (FDA) regulations, the International Conference on Harmonisation (ICH) E6 Guideline for Good Clinical Practice (GCP), and applicable local, state, and federal laws.

Study Assessments: After informed consent is obtained and screening measurements are completed, the patients will return at 4 weeks for injection for primary and secondary efficacy evaluations. Additional evaluations at 6 and 12 weeks will be made in order to determine the duration of effect of Xeomin for secondary efficacy evaluations.

Concomitant therapy includes any prescription or over the counter preparations being taken by the patient at any time from screening through the last study visit. All concomitant medications should be reported to the investigator and recorded.

Patients enrolled in the study will be permitted to take all medication with the exception of the following

* Methylprednisolone within 30 days prior to screening
* Injection of any botulinum toxin within the past 6 months (180days)

During the study patients will be permitted to receive any treatment deemed necessary by the investigator for the management of disease. However patients requiring commencement of excluded therapies will be discontinued from the study and the data will not be used for statistical purposes.

Study Assessments:

Patients must sign informed consent form before any screening evaluations or measurements are performed. Patients must satisfy all of the inclusion criteria and none of the exclusion criteria to be randomized. Information regarding consented patients who are not subsequently randomized will be keep in the regulatory binder.

SAFETY MEASURES

Safety assessments will consist of monitoring and recording adverse events (AE's) and serious adverse events (SAE's). All SAE's will be reported to the FDA Med Watch within 48 business hrs of site notification of such SAE. For this protocol a serious SAE will be defined as any AE that is meets any of the following criteria:

* Fatal (i.e. the AE actually causes or leads to death)
* Life threatening (i.e. the AE in the view of the investigator, placing the patient at immediate risk of death)
* Requires or prolongs hospitalization
* Results in persistent or significant disability/incapacity (i.e. the AE results in substantial disruption to the patients ability to conduct normal life functions)
* A congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product
* Considered a significant medical event by the investigator (e.g, may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above)

The FDA Adverse Event Reporting System Med Watch is a Reporting system for Health Professionals

STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE A detailed description of the statistical methodology will be provided in the statistical analysis plan (SAP) which may deviate from the analysis outlined in the protocol; however, any substantial deviations from the protocol will be detailed in a protocol amendment.

Description of Endpoints

* Primary Endpoint Mean change from injection visit to week 6 in the Modified Ashworth score between Xeomin vs placebo group
* Secondary Endpoints

  * Mean change from injection visit to week 6 in Multiple Sclerosis Impact Scale (MSIS-29) Physical and psychological scores between Xeomin vs placebo group
  * Mean change from injection visit to week 6 in T25FW between Xeomin vs Placebo group.
  * Patient global impression of change (PGIC) between Xeomin vs placebo group
  * Clinical Global Impression of change between Xeomin vs placebo group
  * Mean change from injection visit to week 6 in Likert pain scale between Xeomin vs placebo group
  * Mean change from injection visit to week 6 in MSWS-12 between Xeomin vs placebo group.

Demography and Baseline Disease Characteristics

* Demographic and baseline characteristics will be presented descriptively (i.e., mean, standard deviation, median, range) and analyzed with appropriate statistical methods given the distribution and type of data.

Efficacy

* Analysis Population The Intent-to-Treat population is defined as all subjects who receive at least 1 dose of study treatment and who provide efficacy assessment.
* General Methods of Analysis Descriptive statistics will be provided for all efficacy endpoints. A two-sided test, p-value and confidence interval will be presented for analysis in general.
* Primary Endpoint Analysis The primary endpoint is the mean change from injection visit to week 6 in Modified Ashworth score . A two sample T-test will be used to compare the treatment difference between Xeomin and placebo group. If the data is not normally distributed, Wilcoxon's rank sum test will be used for the analysis.
* Secondary Endpoints Analysis Percent change from injection visit to week 6 will be calculated for the primary endpoint. It will be analyzed similarly as that for the primary endpoint. For secondary endpoints MSIS 29, T25FW, Likert pain scale and MSWS-12 a similar statistical approach as outlined for the primary endpoint will be used to assess the mean changes from injection visit to week 6 in each of the scales between treatment groups.

Patient global impression of change (PGIC) and clinical global Impression of change will be analyzed using the Wilcoxon's rank sum test.

Safety

* Analysis Population The safety population is defined as all subjects who receive at least 1 dose of study treatment.

Adverse events will be listed. Serious AE will be listed as well.

Sample Size Considerations Based on observational study, patients using Xeomin had an improvement of 50% on the Ashworth scale. A sample size of 15 patients per group will provide 80% power to detect a treatment difference of 50% with a 0.05 two-sided significance level using a chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with clinically definite MS, either RRMS or a progressive form (SPMS, PPSM, PRMS)
* Ages 18-65 years.
* Patients must be in a stable state, with no clinical relapses or methylprednisolone treatments in the last 30 days, or have slowly progressive MS, with an EDSS score of 2.0-6.5.
* Patients must have functionally significant spasticity in predominantly one lower extremity as determined by a score of >2 on the Modified Ashworth Scale at screen

Exclusion Criteria:

* Unstable medical or neurological disease
* Known sensitivity to Xeomin
* Prior injection with any botulinum toxin within 6 months
* EDSS score of 7.0 or greater
* Exacerbation of MS within the past 30 days
* Significant cognitive impairment or psychiatric disease
* Advanced arthritis or any other cause of clinically significant limitation of passive range of motion around any of the joints being assessed in the study.
* Concomitant neurologic conditions causing spasticity or rigidity.
* Has had major surgery within 3 months prior to Screening visit that may affect spasticity assessments such as back, lower leg or knee surgeries.
* Use of medications that could influence muscle tone or any anti-spasticity medications must be stable >90 days prior to screening visit and must remain stable throughout study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01-27 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Mean change from injection visit to week 6 in the Modified Ashworth score between Xeomin vs placebo group | injection visit to week 6

SECONDARY OUTCOMES:
Mean change from injection visit to week 6 in Multiple Sclerosis Walking Scale (MSWS-12) between Xeomin vs placebo group | from injection visit to week 6
Change in Patient Global impression of change between Xeomin vs placebo group | change between week 6 and week 12
Mean change from injection visit to week 6 in Multiple Sclerosis Impact Scale (MSIS-29) physical and psychological scores between Xeomin vs placebo group | injection visit to week 6
Mean change from injection visit to week 6 in Timed 25 Foot Walk (T25FW) between Xeomin vs placebo group | injection visit to week 6
Clinical Global impression of change between Xeomin vs placebo group | change between week 6 and week 12
Mean change from injection visit to week 6 in Likert Pain Scale between Xeomin vs placebo group | injection visit to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, MD, Principal Investigator — MS Center of Northeastern New York
Locations (1):
- Multiple Sclerosis Center of Northeastern New York, Latham, New York, United States

REFERENCES:
- [Background] Moore AP. Botulinum toxin A (BoNT-A) for spasticity in adults. What is the evidence? Eur J Neurol. 2002 May;9 Suppl 1:42-7; dicussion 53-61. doi: 10.1046/j.1468-1331.2002.0090s1042.x. PMID 11918649
- [Result] Hesse S, Lucke D, Malezic M, Bertelt C, Friedrich H, Gregoric M, Mauritz KH. Botulinum toxin treatment for lower limb extensor spasticity in chronic hemiparetic patients. J Neurol Neurosurg Psychiatry. 1994 Nov;57(11):1321-4. doi: 10.1136/jnnp.57.11.1321. PMID 7964805
- [Result] Gilmartin R, Bruce D, Storrs BB, Abbott R, Krach L, Ward J, Bloom K, Brooks WH, Johnson DL, Madsen JR, McLaughlin JF, Nadell J. Intrathecal baclofen for management of spastic cerebral palsy: multicenter trial. J Child Neurol. 2000 Feb;15(2):71-7. doi: 10.1177/088307380001500201. PMID 10695888
- [Result] Levin AB, Sperling KB. Complications associated with infusion pumps implanted for spasticity. Stereotact Funct Neurosurg. 1995;65(1-4):147-51. doi: 10.1159/000098887. PMID 8916345
- [Result] Loubser PG, Narayan RK, Sandin KJ, Donovan WH, Russell KD. Continuous infusion of intrathecal baclofen: long-term effects on spasticity in spinal cord injury. Paraplegia. 1991 Jan;29(1):48-64. doi: 10.1038/sc.1991.7. PMID 2023770
- [Result] de Paiva A, Meunier FA, Molgo J, Aoki KR, Dolly JO. Functional repair of motor endplates after botulinum neurotoxin type A poisoning: biphasic switch of synaptic activity between nerve sprouts and their parent terminals. Proc Natl Acad Sci U S A. 1999 Mar 16;96(6):3200-5. doi: 10.1073/pnas.96.6.3200. PMID 10077661
- [Result] Koman LA, Mooney JF 3rd, Smith BP, Walker F, Leon JM. Botulinum toxin type A neuromuscular blockade in the treatment of lower extremity spasticity in cerebral palsy: a randomized, double-blind, placebo-controlled trial. BOTOX Study Group. J Pediatr Orthop. 2000 Jan-Feb;20(1):108-15. PMID 10641699
- [Result] Brashear A, Gordon MF, Elovic E, Kassicieh VD, Marciniak C, Do M, Lee CH, Jenkins S, Turkel C; Botox Post-Stroke Spasticity Study Group. Intramuscular injection of botulinum toxin for the treatment of wrist and finger spasticity after a stroke. N Engl J Med. 2002 Aug 8;347(6):395-400. doi: 10.1056/NEJMoa011892. PMID 12167681
- [Result] Dykstra DD, Sidi AA. Treatment of detrusor-sphincter dyssynergia with botulinum A toxin: a double-blind study. Arch Phys Med Rehabil. 1990 Jan;71(1):24-6. PMID 2297305
- [Result] Yablon SA, Agana BT, Ivanhoe CB, Boake C. Botulinum toxin in severe upper extremity spasticity among patients with traumatic brain injury: an open-labeled trial. Neurology. 1996 Oct;47(4):939-44. doi: 10.1212/wnl.47.4.939. PMID 8857723
- [Result] Snow BJ, Tsui JK, Bhatt MH, Varelas M, Hashimoto SA, Calne DB. Treatment of spasticity with botulinum toxin: a double-blind study. Ann Neurol. 1990 Oct;28(4):512-5. doi: 10.1002/ana.410280407. PMID 2252363
- [Result] Hyman N, Barnes M, Bhakta B, Cozens A, Bakheit M, Kreczy-Kleedorfer B, Poewe W, Wissel J, Bain P, Glickman S, Sayer A, Richardson A, Dott C. Botulinum toxin (Dysport) treatment of hip adductor spasticity in multiple sclerosis: a prospective, randomised, double blind, placebo controlled, dose ranging study. J Neurol Neurosurg Psychiatry. 2000 Jun;68(6):707-12. doi: 10.1136/jnnp.68.6.707. PMID 10811692
- [Result] Borg-Stein J, Pine ZM, Miller JR, Brin MF. Botulinum toxin for the treatment of spasticity in multiple sclerosis. New observations. Am J Phys Med Rehabil. 1993 Dec;72(6):364-8. PMID 8260129
- [Result] Pierson SH, Katz DI, Tarsy D. Botulinum toxin A in the treatment of spasticity: functional implications and patient selection. Arch Phys Med Rehabil. 1996 Jul;77(7):717-21. doi: 10.1016/s0003-9993(96)90015-5. PMID 8670002
- [Result] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714